CLINICAL TRIAL: NCT02629692
Title: A Two-Part Phase 1/2 Study to Determine Safety, Tolerability, Pharmacokinetics, and Activity of K0706, a Novel Tyrosine Kinase Inhibitor (TKI), in Healthy Subjects and in Subjects With Chronic Myeloid Leukemia (CML) or Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia (Ph+ ALL)
Brief Title: Safety and Anti-leukemic Activity of Vodobatinib (K0706) for Treatment of Ph+ CML Resistant/Intolerant to ≥3 Prior CML Therapies
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Pharma Advanced Research Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLR_15_03 V 12 Amendment 12
Record Dates: First submitted 2015-12-10; First posted 2015-12-14 (Estimated); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Healthy (For Part A); Chronic Myeloid Leukemia (for Part B and C)
Keywords: CML; Chronic Myelogenous Leukemia; K0706; Vodobatinib; ponatinib-refractory/intolerant; treatment refractory chronic myeloid leukemia; Ponatinib
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Capsules

STUDY DESIGN:
Intervention Model Description: Part A: Single ascending dose in healthy volunteers.
  Part B: Multiple ascending dose safety and tolerability study in subjects with CML or Ph + ALL.
  Part C: Efficacy and safety study in subjects with treatment-resistant CML
Masking Description: Part B and C: Single arm (Open-label)
  Part A: 2 arms: Investigational agent arm and Placebo arm (Double-blind).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vodobatinib (K0706) capsules (Experimental)
  Interventions: Drug: Vodobatinib (K0706) capsules

INTERVENTIONS:
Drug: Vodobatinib (K0706) capsules — Part A: Vodobatinib (K0706) capsules in single ascending doses.
  Part B: Oral Vodobatinib (K0706) capsules in multiple ascending doses, once daily.
  Part C: Oral Vodobatinib (K0706) capsules at recommended phase 2 dose of 174 mg, once daily.

SUMMARY:
Phase 1/2 study to determine safety, tolerability, pharmacokinetics, and anti-leukemic activity of Vodobatinib (K0706) in treatment-refractory/intolerant CML

DETAILED DESCRIPTION:
Part A ( for Healthy volunteers) of the study is completed.

Part B dose-escalation study is completed. Recruitment in dose expansion is completed.

Part C study in subjects with treatment-resistant/intolerant is ongoing for the enrolled subjects.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written, and dated, informed consent
* Male or female aged ≥ 18 years
* Willing and able to comply with the scheduled visits
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Subjects diagnosed with Ph+ CML-CP, Ph+ CML-AP, Ph+ CML-BP, who are resistant and/or intolerant to ≥ 3 prior TKIs one of which includes ponatinib (Part C).

Exclusion Criteria:

* Presence of T315I (PART C)
* Any major surgery, as determined by the Investigator, within 4 weeks of IMP administration
* Inability to undergo venipuncture and/or tolerate venous access
* Positive exclusion tests: urine pregnancy tests (if applicable), HIV, hepatitis B surface antigen, or hepatitis C virus
* Known or suspected history of significant drug abuse as judged by the Investigator
* Received any other investigational agent within 30 days or a washout of at least 5 half-lives, whichever is longer of IMP administration
* Subjects who are eligible for potentially curative therapy that is available, including hematopoietic stem cell transplant
* Another primary malignancy within the past 3 years or earlier (except for adequately treated non-melanoma skin cancer or cervical cancer in situ

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2016-06-27 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
To determine the Maximum Tolerated Dose (MTD) as determined by frequency of Dose Limiting Toxicities | Dose Limiting toxicities observed over a 4 week period
  PART B
Incidence and severity of treatment emergent AEs as assessed by CTCAE v4.03 | All subjects will be followed up for 60 months from the first dose of Vodobatinib (K0706)
  PART B
For CML subjects in CP at study entry | All subjects will be followed up for 60 months from the first dose of Vodobatinib (K0706)
  PART C: Proportion of subjects achieving Major Cytogenetic Response [ defined as complete cytogenetic response (CCyR; 0% Ph+metaphases) or partial cytogenetic response (PCyR; 1-35% Ph+ metaphases)] as assessed by conventional Karyotyping of Bone marrow aspirate
For CML subjects in AP at study entry | All subjects will be followed up for 60 months from the first dose of Vodobatinib (K0706)
  PART C: Proportion of subjects achieving Major Hematologic Response [ defined as complete hematologic response (CHR) or no evidence of leukemia (NEL)] as assessed by complete blood count of peripheral blood sample
For CML subjects in BP at study entry | All subjects will be followed up for 60 months from the first dose of Vodobatinib (K0706)
  PART C: Proportion of subjects achieving Major Hematologic Response [defined as complete hematologic response (CHR) or no evidence of leukemia (NEL)] as assessed by complete blood count of peripheral blood sample

SECONDARY OUTCOMES:
Pharmacokinetic profile of K0706 - Cmax [The maximum (peak) observed drug concentration after dose administration] | All subjects will be followed for up to approximately 60 months after the first dose of Vodobatinib (K0706)
  PART B and PART C
Pharmacokinetic profile of Vodobatinib (K0706) - Tmax [The time to reach maximum (peak) drug concentration after dose administration] | All subjects will be followed for up to approximately 60 months after the first dose of Vodobatinib (K0706)
  PART B and PART C
Pharmacokinetic profile of Vodobatinib (K0706) - Cmin [ Minimum observed drug concentration after dose administration] | All subjects will be followed for up to approximately 60 months after the first dose of Vodobatinib (K0706)
  PART B and PART C
In subjects with CML- CP:Proportion of subjects achieving Complete Hematological Response as assessed by complete blood count of peripheral blood sample | All subjects will be followed up for 60 months from the first dose of Vodobatinib (K0706)
  PART C
In subjects with CML- CP:Proportion of subjects achieving Complete Cytogenetic Response as assessed by conventional Karyotyping of Bone marrow aspirate | All subjects will be followed up for 60 months from the first dose of Vodobatinib (K0706)
  PART C
In subjects with CML- CP:Proportion of subjects achieving Major Molecular Response as assessed by BCR-ABL transcript levels (BCR-ABL1 ratio of ≤ 0.1%) in peripheral blood using PCR (Polymerase Chain Reaction) | All subjects will be followed up for 60 months from the first dose of Vodobatinib (K0706)
  PART C
In subjects with CML-AP & BP: Proportion of subjects achieving Complete cytogenetic response as assessed by conventional Karyotyping of Bone marrow aspirate | All subjects will be followed up for 60 months from the first dose of Vodobatinib (K0706)
  PART C
In subjects with CML-AP & BP: Proportion of subjects achieving Partial Cytogenetic Response (PCyR) as assessed by conventional Karyotyping of Bone marrow aspirate | All subjects will be followed up for 60 months from the first dose of K0706
  Part C
In subjects with CML-AP & BP: Proportion of subjects achieving Major Molecular Response as assessed by BCR-ABL transcript levels (BCR-ABL1 ratio of ≤ 0.1%) in peripheral blood using PCR (Polymerase Chain Reaction) | All subjects will be followed up for 60 months from the first dose of Vodobatinib (K0706)
  PART C
Time to Major Cytogenetic Response (MCyR): Time to MCyR is the time from first dose to first MCyR (0-35% Ph+ metaphases) ; computed only for subjects who achieved MCyR | All subjects will be followed up for 60 months from the first dose of Vodobatinib (K0706)
  PART C
Time to Major Molecular Response : Time to MMR is the time from first dose to first MMR (BCR-ABL1 ratio of ≤ 0.1%) computed only for subjects who achieved MMR | All subjects will be followed up for 60 months from the first dose of Vodobatinib (K0706)
  PART C
In all subjects Progression free survival (PFS) | All subjects will be followed up for 60 months from the first dose of Vodobatinib (K0706)
  PART C
In all subjects Overall survival (OS) | All subjects will be followed up for 60 months from the first dose of Vodobatinib (K0706)
  PART C
Incidence and severity of treatment emergent AEs as assessed by CTCAE v5.0 | All subjects will be followed up for 60 months from the first dose of Vodobatinib (K0706)
  PART C

CONTACTS AND LOCATIONS:
Locations (37):
- United States (8):
  - The Oncology Institute of Hope and Innovation, Innovative Clinical Research Institute, Downey, California
  - UCLA Hematologic Malignancy Program, Los Angeles, California
  - Mayo Clinic, Jacksonville, Florida
  - Board of Regents of the University System of Georgia, Augusta, Georgia
  - Memorial Sloan Kettering Cancer Center - MAIN, New York, New York
  - Baylor University Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute University of Utah, Salt Lake City, Utah
- Cliniques Universitaires Saint-Luc, Brussels, Belgium
- France (3):
  - Institut Paoli Calmettes, Marseille, Bouches-du-Rhône
  - Centre Léon Bérard, Lyon, Rhone
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Rhone
- Debreceni Egyetem, Debrecen, Hungary
- India (5):
  - Prince Aly Khan Hospital, Mumbai, Maharashtra
  - Tata Memorial Hospital, Mumbai, Maharashtra
  - Sahyadri Specialty Hospital, Pune, Maharashtra
  - Meenakshi Mission Hospital & Research Centre, Madurai, Tamil Nadu
  - Tata Medical Centre, Kolkata, West Bengal
- Italy (5):
  - Istituto Scientifico Romagnolo Per Lo Studio e La Cura Dei Tumori, Meldola, Forli - Cesena
  - Azienda Socio Sanitaria Territoriale di Monza (Presidio San Gerardo), Monza, Milano
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale Sant'Eugenio, Roma
  - Azienda Ospedaliera Universitaria Policlinico Umberto I - Università di Roma La Sapienza, Roma
- Romania (3):
  - Spitalul Clinic Colentina, Bucharest
  - Institutul Oncologic "Prof. Dr. Ion Chiricuta" Cluj-Napoca, Cluj-Napoca
  - Spitalul Clinic Municipal Filantropia Craiova, Craiova
- South Korea (2):
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul, Gyeonggi-do
  - Uijeongbu Eulji Medical Center, Eulji University, Gyeonggi-do
- Spain (5):
  - ICO Badalona - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
- Turkey (Türkiye) (2):
  - Hacettepe University Hospital, Altındağ
  - Kayseri Erciyes University Hospital, Kayseri
- United Kingdom (2):
  - King's College Hospital, London, Greater London
  - Hammersmith Hospital, London, Greater London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cortes JE, Kim DW, Saikia T, Khattry N, Rathnam K, Alvarado Y, Hannah G, Tantravahi SK, Apperley JF, Charbonnier A, Garcia-Gutierrez V, Lucchesi A, Dima D, Illes A, Popov VM, Abruzzese E, Nag A, Apte S, Badar T, Yao SL, Saxena U, Sreenivasan J, Inamdar S, Chimote G, Nicolini FE. Vodobatinib for patients with Philadelphia chromosome-positive chronic myeloid leukaemia resistant or intolerant to multiple lines of previous therapy: an open-label, multicentre, phase 1/2 trial. Lancet Haematol. 2025 Mar;12(3):e201-e213. doi: 10.1016/S2352-3026(24)00354-5. Epub 2025 Feb 7. PMID 39929221